CLINICAL TRIAL: NCT03452540
Title: A Randomised, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Efficacy and Safety of Orally Administered DS102 in Patients With Acute Decompensated Alcoholic Hepatitis.
Brief Title: Efficacy and Safety of Orally Administered DS102 in Patients With Acute Alcoholic Hepatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Afimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS102A-05-AH1; 2018-000819-25 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Severe Acute Decompensated Alcoholic Hepatitis
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1000mg DS102 (BID) (Experimental): Participants assigned to the open label pilot phase received 1000mg DS102 (BID)for 28 days.
  Interventions: Drug: 1000mg DS102 (BID)

INTERVENTIONS:
Drug: 1000mg DS102 (BID) — Participants assigned to the open label pilot phase received 1000mg DS102 (BID)for 28 days.

SUMMARY:
The purpose of this randomised, double-blind, placebo-controlled, phase II study is to assess the efficacy and safety of orally administered DS102 in adult patients with acute decompensated alcoholic hepatitis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years and older
2. Total bilirubin of ≥ 5 mg/dl (85μmol/l)
3. Patients with definite or probable AH
4. MELD ≥18 at baseline visit
5. MDF ≥32 at baseline visit
6. AST ≥50 U/L
7. AST':ALT ratio > 1.5
8. Female patients, or female partners of male patients, of child bearing potential must use highly effective birth control methods or have a sterilised partner for the duration of the study. Highly effective birth control methods are defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include intrauterine device or sexual abstinence.

   Note: A woman is considered of child bearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy Note: Hormonal contraceptives are contraindicated in patients with severe hepatic diseases and are not acceptable as a birth control method in this study Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject
9. Patient and/or legally authorised representative must provide informed consent
10. Able to swallow the provided study medication
11. Not eligible for liver transplant during this hospitalisation

Exclusion Criteria:

1. Pregnant or lactating females.
2. Spontaneous liver function improvement defined by decrease of bilirubin level and MDF of >10% within 5 days of hospital admission
3. Grade 4 hepatic encephalopathy (West Haven Criteria)
4. Type 1 hepatorenal syndrome (HRS) or a serum creatinine >2 x ULN or the requirement for haemodialysis
5. History of hypersensitivity to any substance in DS102 capsules or placebo capsules.
6. Alcohol abstinence of >6 weeks prior to screening
7. Duration of clinically apparent jaundice >3 months prior to baseline
8. Other causes of liver disease including:

   1. Evidence of chronic viral hepatitis (Hepatitis B DNA positive or HCV RNA positive)
   2. Biliary obstruction
   3. Hepatocellular carcinoma
   4. Wilsons disease
   5. Budd Chiari Syndrome
   6. Non-alcoholic fatty liver disease
9. History of or active non-liver malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas).
10. Previous entry into the study
11. AST >400 U/L or ALT >270 U/L
12. Treatment with any experimental drug within 30 days prior to Day 0 visit (Baseline), or 5 half-lives (whichever is longer).
13. Patients who have used dietary supplements rich in omega-3 or omega-6 fatty acids in the four weeks prior to baseline.
14. Patients dependent on inotropic support (adrenaline or noradrenaline), including Terlipressin
15. Active variceal haemorrhage on this admission requiring more than 2 units of blood to maintain haemoglobin level within 48 hours
16. Presence of refractory ascites
17. Untreated or unresolved sepsis
18. Patients with cerebral haemorrhage, extensive retinal haemorrhage, acute myocardial infarction (within last 6 weeks) or severe cardiac arrhythmias (not including atrial fibrillation)
19. Known infection with HIV at screening.
20. Significant systemic or major illnesses other than liver disease that, in the opinion of the investigator, would preclude or interfere with treatment with DS102 and/or adequate follow up.
21. Previous liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thursz, Principal Investigator — Imperial College London
Locations (8):
- United States (6):
  - Schiff Center for Liver Diseases (University Hospital Miami), Miami, Florida
  - Cleveland Clinic Florida, Miami, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours Liver Institute of Richmond and Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
- Georgia (2):
  - Batumi Referral Hospital, Batumi
  - Saint Nikolozi Surgery Center, Kutaisi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre, double blind, placebo controlled, 2-arm parallel group comparison (Phase 2) study, preceded by an open label pilot phase, in which six patients were to receive open label treatment with 2000mg DS102 (1000mg BID) within 30 minutes after a meal for 28 days.
Pre-assignment Details: A total of 126 participants were planned with actual enrolment in the study. 9 participants completed the open label pilot phase before the study was ended prematurely due to futility purposes.
Period: Overall Study
Arm/Group | 1000mg DS102 (BID)
Started | 9
Completed | 5
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other SAE and AE | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all patients who received at least one dose of investigational product. Patients were analysed according to the treatment they were assigned to, irrespective of what treatment they actually received.
Arm/Group | 1000mg DS102 (BID)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and SUSARs.
Description: To evaluate the safety of orally administered DS102 in the treatment of adult patients with severe acute decompensated AH.
Time Frame: Up to 28 days.
Population: as for baseline characteristics
Measure: Number; unit: Number of Events
Arm/Group | 1000mg DS102 (BID)
Number analyzed (Participants) | 9
Number of Events
  Total Number of TEAEs | 7
  Total Number of Serious TEAEs | 4
  Total Number of Serious Treatment Related TEAEs | 1
  Total Number of Treatment Related TEAEs | 1
  Total Number of Not Treatment Related TEAEs | 6

2. Primary Outcome: Descriptive Statistics for Plasma Total 15(S)-HEPE and Unesterified 15(S)-HEPE Pharmacokinetic Results for 1000 mg BD DS102 Administered Orally Twice-daily to Patients With Alcoholic Hepatitis
Description: Descriptive Statistics for Plasma Total 15(S)-HEPE and Unesterified 15(S)-HEPE Pharmacokinetic Results for 1000 mg BD DS102 Administered Orally Twice-daily to Patients with Alcoholic Hepatitis.
Time Frame: Up to 7 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1000mg DS102 (BID)
Number analyzed (Participants) | 9
ng/mL
  Day 0 Unesterified 15(S)-HEPE | 542 (399.4)
  Day 7 Unesterified 15(S)-HEPE | 1060 (1073)
  Day 0 Total 15(S)-HEPE | 3110 (3721)
  Day 7 Total 15(S)-HEPE | 4470 (3601)

ADVERSE EVENTS:
Time Frame: Up to 90 days.
Description: An adverse event is any undesirable experience occurring to a patient that has signed the ICF and who has taken their first dose of the study drug, whether or not considered related to the investigational medicinal product (IMP). All Adverse Events (AEs) were recorded in the CRF, defining relationship to IMP and severity.
Arm/Group | 1000mg DS102 (BID)
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000mg DS102 (BID) (N=9)
Cardiac Arrest (Cardiac disorders) | 1
Septic Shock (Infections and infestations) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Mental status change (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000mg DS102 (BID) (N=9)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Localised Oedema (General disorders) | 1
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Aspartate Aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood Alkaline phosphate increased (Investigations) | 1
Paracentesis (Investigations) | 1
Palpitations (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Head Injury (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
Confusional State (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination - The study was stopped at the end of the pilot phase (n=9) as the sponsor prioritised other therapeutic indications, so no patients were enrolled in the double-blind phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03452540/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03452540/SAP_001.pdf